CLINICAL TRIAL: NCT01316601
Title: A Study to Assess Efficacy, Safety and Tolerability of the Anti-IL-13 Monoclonal Antibody QAX576 in the Treatment of Perinanal Fistulas in Patients Suffering From Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerhard Rogler (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Gerhard Rogler, Prof.Dr.Dr. Gerhard Rogler, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Novartis CQAX576
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: QAX567

SUMMARY:
Test safety and efficacy and of a novel IL-13 AB in the treatment of perianal fistulas

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: - diagnosis of Crohn's disease > 6 month with fistula - at least 1 ineffective fistula treatment in the past

Exclusion criteria: - TNF a antibody treatment failed in the past

- planned surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
complete closure of fistula

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland